CLINICAL TRIAL: NCT07367035
Title: The Effect of an Art-Based Emotion Regulation Program on Anxiety, Emotion Regulation Skills, and Symptom Burden in Adolescents Undergoing Cancer Treatment: A Randomized Controlled Trial
Brief Title: Art-Based Emotion Regulation Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Hazal Ozdemir Koyu, Dr. Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2026-64
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Children With Cancer
Keywords: Adolescent Cancer; Pediatric Oncology; Art-Based Intervention; Emotion Regulation; Anxiety; Symptom Burden
MeSH Terms: conditions — Emotional Regulation; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is designed as a single-blind, parallel-group randomized controlled trial. Participants will be allocated in a 1:1 ratio to either the intervention group or the control group using stratified block randomization based on age and gender. The intervention group will receive an art-based emotion regulation program in addition to routine care, while the control group will receive routine care alone. There will be no crossover between groups, and outcome assessments will be conducted at baseline and at the end of the 4-week intervention period.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the art-based intervention, blinding of participants and intervention providers is not feasible. However, outcome assessors will be blinded to group allocation. Data collection and outcome assessments will be conducted by assessors who are not involved in the intervention delivery and are unaware of participants' group assignments to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Received Standart Care
- rt-Based Emotion Regulation Program (Experimental): Received Art-Based Emotion Regulation Program
  Interventions: Other: Art-Based Emotion Regulation Program

INTERVENTIONS:
Other: Art-Based Emotion Regulation Program — The Art-Based Emotion Regulation Program is a structured, non-pharmacological intervention designed to support emotional regulation and reduce anxiety and symptom burden in adolescents undergoing cancer treatment. The program is delivered over a 4-week period and combines relaxation techniques with expressive art-based activities.
  The intervention includes progressive muscle relaxation exercises, emotion-color mapping activities, and gratitude mandala practices. During the first week, participants receive a guided progressive muscle relaxation exercise delivered via video, with the initial session conducted together with the researcher. Participants are then instructed to practice the relaxation exercise at least twice per week throughout the intervention period.
  Emotion-color mapping activities are conducted during weeks 1 to 3, allowing adolescents to visually express emotions and treatment-related symptoms using colors and drawings. Changes in emotional states and symptom intensit
  Arms: rt-Based Emotion Regulation Program

SUMMARY:
Adolescents receiving cancer treatment often experience increased anxiety, difficulties in emotion regulation, and a high symptom burden due to treatment-related physical effects and psychosocial stressors. Supportive, non-pharmacological interventions that promote emotional regulation are therefore needed.

The purpose of this randomized controlled trial is to evaluate the effect of an art-based emotion regulation program on anxiety levels, emotion regulation skills, and symptom burden in adolescents undergoing cancer treatment.

This single-blind, parallel-group randomized controlled study will include 60 adolescents aged 10-18 years receiving cancer treatment at Gazi University Health Application and Research Center and Etlik City Hospital Pediatric Hematology-Oncology units between January 30, 2026 and March 20, 2027. Participants will be randomly assigned to either the intervention group or the control group. The intervention group will receive a 4-week art-based emotion regulation program, while the control group will receive routine care. Outcomes will be assessed using validated self-report measures at baseline and at the end of the intervention period.

DETAILED DESCRIPTION:
Adolescents undergoing cancer treatment frequently experience a combination of physical symptoms and psychosocial stressors that negatively affect their emotional well-being, anxiety levels, and ability to regulate emotions. Difficulties in emotion regulation may intensify perceived symptom burden and interfere with treatment adherence and overall quality of life. Art-based interventions offer developmentally appropriate, expressive, and non-invasive strategies to support emotional regulation in this population.

This study is designed as a single-blind, parallel-group randomized controlled trial to examine the effectiveness of an art-based emotion regulation program in adolescents receiving cancer treatment. The study will be conducted between January 30, 2026 and March30, 2027 at the Pediatric Hematology-Oncology units of Gazi University Health Application and Research Center and Etlik City Hospital.

A total of 60 adolescents aged 10-18 years who have been receiving cancer treatment for at least six months will be enrolled and randomly assigned to either the intervention group (n=30) or the control group (n=30). Stratified block randomization based on age and gender will be performed by an independent statistician using an online randomization tool. Outcome assessors will be blinded to group allocation.

The intervention group will participate in a 4-week art-based emotion regulation program consisting of progressive muscle relaxation exercises, emotion-color mapping activities, and gratitude mandala practices. During the first week, adolescents will receive a progressive muscle relaxation video and complete the first session together with the researcher. They will then be asked to practice the exercise at least twice weekly throughout the program. Emotion-color mapping activities will be conducted during weeks 1-3 to help adolescents visually express and monitor changes in emotional states and symptom intensity. In the second week, a gratitude mandala activity will be added to enhance awareness of positive emotions. Weekly follow-up discussions will be conducted to support engagement and reflection. In the fourth week, relaxation exercises will continue, emotion-color maps will be reviewed for change, and post-test assessments will be completed.

The control group will receive routine hospital care without any additional intervention. Both groups will complete the same assessment tools at baseline and at the end of the fourth week.

Primary and secondary outcomes will be measured using the State Anxiety Inventory for Children, the Emotion Regulation Questionnaire for Children and Adolescents, and the Pediatric Symptom Screening Tool (SSPedi). The findings of this study are expected to provide evidence for the effectiveness of art-based emotion regulation interventions as a supportive, feasible, and non-pharmacological approach in adolescent oncology care.

ELIGIBILITY:
* Inclusion Criteria for the Study:

  1. Receiving cancer treatment for at least 6 months,
  2. Aged between 10 and 18 years,
  3. The participant and their parent/guardian consent to participate in the study and provide written informed consent.

Exclusion Criteria:

1. Those who have experienced a significant life event (death, relocation, etc.) unrelated to their illness in the last six months,
2. Those who have not received chemotherapy treatment,
3. Those in the terminal stage,
4. Those with a severe psychological diagnosis and taking medication

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Inventory for Children (SAIC) | Baseline (pre-intervention) and immediately post-intervention (at the end of the 4-week intervention period).
  The State Anxiety Inventory for Children (SAIC) was developed by Spielberger (1973) to assess situational anxiety levels in children and adolescents. The Turkish validity and reliability study was conducted by Özusta (1995). The scale consists of 40 items, including 20 items measuring state anxiety and 20 items measuring trait anxiety. In this study, only the State Anxiety subscale is used to evaluate the child's current feelings of anxiety. Total scores range from 20 to 60, with higher scores indicating higher anxiety levels. The original scale demonstrated Cronbach's alpha values between 0.78 and 0.81, while the Turkish version reported a Cronbach's alpha of 0.82 for the state anxiety subscale. The scale has been widely used among children and adolescents aged 9-18 years in Turkey.
Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA) | Baseline (pre-intervention) and immediately post-intervention (at the end of the 4-week intervention period).
  The Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA) was originally developed by Gullone and Taffe (2012) and adapted into Turkish by Tetik and Önder (2021). The scale is a self-report measure designed to assess differences in emotion regulation strategies among children aged 10-18 years. It consists of 10 items and includes two subscales: Cognitive Reappraisal (6 items) and Expressive Suppression (4 items). Items are rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate more frequent use of the corresponding emotion regulation strategy. The Turkish version demonstrated good internal consistency, with Cronbach's alpha values of 0.83 for the reappraisal subscale and 0.75 for the suppression subscale.
Symptom Screening in Pediatrics Tool (SSPedi) | Baseline (pre-intervention) and immediately post-intervention (at the end of the 4-week intervention period).
  The Symptom Screening in Pediatrics Tool (SSPedi) is a validated instrument developed to assess symptom burden in children aged 8-18 years undergoing cancer treatment. The original validity and reliability study for the electronic version was conducted by O'Sullivan et al. (2018), reporting a Cronbach's alpha coefficient of 0.88. The tool evaluates 15 common symptoms experienced by children over the past two days, with each symptom rated using a 5-point Likert scale. Total scores range from 0 to 60, with higher scores indicating greater symptom burden and distress. The Turkish validity and reliability study was conducted by Çelik et al. (2021).

IPD SHARING:
Plan to Share IPD: Undecided
Researchers who provide a methodologically sound proposal may request access to the data. Requests will be reviewed by the principal investigator. Data will be shared for scientific research purposes only and after approval of a data use agreement.

REFERENCES:
- [Result] 1. Kisecik Sengul, Z., & Kilicarslan, E. (2025). Investigation into the impact of technology-based motivation program applied to children following cancer diagnosis and their families: a randomized controlled study. BMC psychology, 13(1), 857. 2. Lewandowska, A., Lewandowski, T., Bartosiewicz, A., Papp, K., Zrubcová, D., Šupínová, M., Stryjkowska-Góra, A., Laskowska, B., Joniec, G., & Apay, S. E. (2024). Prevalence of Anxiety and Depression among Parents of Children with Cancer-A Preliminary Study. Children, 11(10), 1227. 3. O'Sullivan, C., Dupuis, L. L., Gibson, P., Johnston, D. L., Baggott, C., Portwine, C., Spiegler, B., Kuczynski, S., Tomlinson, D., & Tomlinson, G. A. (2018). Evaluation of the electronic self-report Symptom Screening in Pediatrics Tool (SSPedi). BMJ supportive & palliative care, 8(1), 110-116. 4. Oner, N. and LeCompte, A. (1983). Durumluluk surekli kaygi envanteri el kitabi (The handbook of the state-trait anxiety inventory. In: Istanbul: Bogazici 5. Çelik, R., Törüner, E. K., Altay, N., & Bayram, D. (2024). The Validity-Reliability Study of Turkish Version of Electronical Symptom Screening Tool (8-18) in SSPedi-Pediatric Patients with Cancer. Clinical and Experimental Health Sciences, 14(3), 827-834 6. Özmen, D., Özmen, E., Çetinkaya, A., & Akil, I. Ö. (2016). Ergenlerde sürekli öfke ve öfke ifade tarzları. Anatolian Journal of Psychiatry/Anadolu Psikiyatri Dergisi, 17(1). 7. Nasıroğlu, S., Yolga Tahiroğlu, A., Avcı, A., Gül Çelik, G., & Öztürk, Z. (2012). İstismara uğramış çocuk ve ergenlerin yatarak tedavisi. Anatolian Journal of Psychiatry/Anadolu Psikiyatri Dergisi, 13(4). 8. Tetik, S., & Önder, F. C. (2021). Çocuk Ve Ergenlerde Duygu Düzenleme Ölçeğinin Türkçeye Uyarlanmasi. Çukurova Üniversitesi Sosyal Bilimler Enstitüsü Dergisi, 30(2), 87-100. 9. Jung, C. G. Mandala symbolism (R. F. C. Hull. Volume 9, Part I, The Collected Works of C. G. Jung). Princeton, NJ: Princeton University Press. 1973, p: 100-380. 10. Bandura, A. (1997). Self-